CLINICAL TRIAL: NCT07086144
Title: Efficacy of a Myocardial Panel (Virological, Bacterial and Autoimmune) in the Management and Treatment of Pediatric Myocarditis Complicated With Arrhythmias or Ventricular Dysfunction
Brief Title: Efficacy of a Myocardial Panel in the Management and Treatment of Pediatric Myocarditis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Principal investigator, Azienda Ospedaliero, Universitaria Ospedali Riuniti
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCPC - SALESI 001/2025
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Myocarditis
Keywords: pediatric myocarditis; Arrhythmias; Myocarditis panel; Etiological therapy; Myocardial dysfunction
MeSH Terms: conditions — Myocarditis; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: 15 patients managed and treated in 2024 without applying the myocarditis panel with 15 patients from 2025, in which management and treatment were driven by the panel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myocarditis Panel (Experimental): N=15 patients from 2025, in which management and treatment of arrhythmias and or myocardial dysfunction were driven by the panel
  Interventions: Diagnostic Test: Determination of viral genome, bacterial serology, and markers of inflammation in pediatrics diagnosed with myocarditis
- No Panel (No Intervention): The 15 patients managed and treated for arrhythmias or myocardial dysfunction in 2024 without applying the myocarditis panel

INTERVENTIONS:
Diagnostic Test: Determination of viral genome, bacterial serology, and markers of inflammation in pediatrics diagnosed with myocarditis — N=15 patients from 2025, in which management and treatment of arrhythmias and or myocardial dysfunction were driven by the panel
  Arms: Myocarditis Panel

SUMMARY:
The goal of this observational study is to determine the efficacy a of combined management and treatment driven by the systematic determination of viral genome, bacterial serology, and markers of inflammation in pediatric patients (< 18 years old) diagnosed with myocarditis complicated by arrhythmias (supraventricular and ventricular tachycardias and heart block) or ventricular dysfunction (left ventricular ejection fraction < 50% or right ventricular fractional area change < 35%).

The main question it aims to answer is: Does this panel help resolve arrhythmias or myocardial dysfunction due to myocarditis during hospitalisation and follow-up?

Researchers will compare patients managed and treated in 2024 without applying the myocarditis panel with those enrolled in 2025 who received the panel. Arrhythmias and myocardial dysfunction will be managed in accordance with recent guidelines. Antiviral, antibiotic or immunosuppressive therapies will be implemented in addition to standard therapy when required by the panel.

DETAILED DESCRIPTION:
The Investigators will enrol consecutive pediatric patients (< 18 years old) presenting with myocarditis complicated by arrhythmias or ventricular dysfunction.

The participants will undergo routine daily visits and electrocardiographic and echocardiographic assessment during hospitalisation (within 8 weeks).

During follow-up, a routine visit including an echocardiogram, ECG, and blood tests (complete blood count, liver function tests, renal function tests, inflammation indices, and myocardial necrosis tests) will be performed within the first 40 days of discharge; thereafter, every 3 months after discharge for a total of 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All the consecutive pediatric patients (< 18 years old) presenting with myocarditis complicated by arrhythmias or myocardial dysfunction

Exclusion Criteria:

* Refused consent to be included in the study given by parents or legal tutors
* Uncomplicated myocarditis presenting without arrhythmias or myocardial dysfunction

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Arrhythmias duration | From enrollment to the end of the hospitalisation (maximum of 8 weeks)
  Total duration of in-hospital arrhythmias assessed by electrocardiography
Myocardial dysfunction | From enrollment to the end of the hospitalisation (maximum of 8 weeks)
  Total duration of myocardial dysfunction assessed by echocardiography

SECONDARY OUTCOMES:
Follow-up | 6 months
  Recurrences of arrhythmias or myocardial dysfunction at the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Francesco Bianco, Ancona, The Marches, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon reasonable requests from other investigators.

REFERENCES:
- [Background] Pompa AG, Beerman LB, Feingold B, Arora G. Electrocardiogram changes in pediatric patients with myocarditis. Am J Emerg Med. 2022 Sep;59:49-53. doi: 10.1016/j.ajem.2022.06.027. Epub 2022 Jun 17. PMID 35779288
- [Background] Law YM, Lal AK, Chen S, Cihakova D, Cooper LT Jr, Deshpande S, Godown J, Grosse-Wortmann L, Robinson JD, Towbin JA; American Heart Association Pediatric Heart Failure and Transplantation Committee of the Council on Lifelong Congenital Heart Disease and Heart Health in the Young and Stroke Council. Diagnosis and Management of Myocarditis in Children: A Scientific Statement From the American Heart Association. Circulation. 2021 Aug 10;144(6):e123-e135. doi: 10.1161/CIR.0000000000001001. Epub 2021 Jul 7. PMID 34229446
- [Background] Dasgupta S, Iannucci G, Mao C, Clabby M, Oster ME. Myocarditis in the pediatric population: A review. Congenit Heart Dis. 2019 Sep;14(5):868-877. doi: 10.1111/chd.12835. Epub 2019 Aug 21. PMID 31432626
- [Background] Ammirati E, Veronese G, Bottiroli M, Wang DW, Cipriani M, Garascia A, Pedrotti P, Adler ED, Frigerio M. Update on acute myocarditis. Trends Cardiovasc Med. 2021 Aug;31(6):370-379. doi: 10.1016/j.tcm.2020.05.008. Epub 2020 Jun 1. PMID 32497572
- [Background] Ammirati E, Moslehi JJ. Diagnosis and Treatment of Acute Myocarditis: A Review. JAMA. 2023 Apr 4;329(13):1098-1113. doi: 10.1001/jama.2023.3371. PMID 37014337
- [Background] Ammirati E, Frigerio M, Adler ED, Basso C, Birnie DH, Brambatti M, Friedrich MG, Klingel K, Lehtonen J, Moslehi JJ, Pedrotti P, Rimoldi OE, Schultheiss HP, Tschope C, Cooper LT Jr, Camici PG. Management of Acute Myocarditis and Chronic Inflammatory Cardiomyopathy: An Expert Consensus Document. Circ Heart Fail. 2020 Nov;13(11):e007405. doi: 10.1161/CIRCHEARTFAILURE.120.007405. Epub 2020 Nov 12. PMID 33176455